CLINICAL TRIAL: NCT03961360
Title: Effectiveness of Higher Aspirin Dosing for Prevention of Preeclampsia in High Risk Obese Gravida: An Open Label, Comparative Effectiveness, Randomized Controlled Trial (ASPREO Trial)
Brief Title: Effectiveness of Higher Aspirin Dosing for Prevention of Preeclampsia in High Risk Obese Gravida
Acronym: ASPREO
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Farah Hassan Amro, Clinical Fellow OBGYN, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HSC-MS-18-1073
Record Dates: First submitted 2019-04-16; First posted 2019-05-23 (Actual); Results first posted 2024-05-08 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-04

CONDITIONS: Pre-Eclampsia; Hypertension in Pregnancy; Obesity
MeSH Terms: conditions — Pre-Eclampsia; Hypertension, Pregnancy-Induced; Obesity | interventions — Aspirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- 162 mg/day Aspirin (Experimental)
  Interventions: Drug: Aspirin 162 mg
- 81 mg/day Aspirin (Active Comparator)
  Interventions: Drug: Aspirin 81 mg

INTERVENTIONS:
Drug: Aspirin 81 mg — Low dose aspirin was initially reported as having a beneficial effect at preeclampsia
  Arms: 81 mg/day Aspirin
Drug: Aspirin 162 mg — Low dose aspirin was initially reported as having a beneficial effect at preeclampsia
  Arms: 162 mg/day Aspirin

SUMMARY:
To compare the incidence of preeclampsia in obese pregnant women (BMI greater than 30) with a singleton gestation at less than 20 weeks and either a history of preeclampsia in a prior pregnancy or stage I hypertension or pre-gestational diabetes who are randomized to either 81mg/day aspirin or 162mg/day aspirin.

ELIGIBILITY:
Inclusion Criteria

* A singleton gestation at less than 20 weeks at time of enrollment, with a BMI greater than or equal to 30 and one of the following:

  1. History of preeclampsia in a prior pregnancy
* Diagnosis will be obtained by review of records, and if unavailable then patient history. Preeclampsia diagnosis may be made in antepartum or postpartum period.

OR 2. At least stage I hypertension during pregnancy

* Stage I hypertension is defined as a systolic blood pressure between 130- 139 mm Hg or diastolic blood pressure between 80-89 mm Hg21
* This blood pressure criteria is met regardless of medication usage
* The patient must have a blood pressure reading ≥ 130-139/80-89 mm Hg at least during 1 clinic visit during the current pregnancy; before or at time of enrollment

OR

3. Pre-gestational diabetes

* Type 1 and Type 2 diabetics are included
* Gestational diabetes mellitus diagnosed prior to 20 weeks gestational age will also be included

Exclusion Criteria

* Known allergy/prior adverse reaction/any medical condition where aspirin is contraindicated
* Already on aspirin prior to pregnancy
* Baseline renal Disease
* Baseline proteinuria identified at time of enrollment, defined as urine analysis with 3+ protein, or urine protein to creatinine ratio ≥ 0.3
* Systemic Lupus Erythematosus
* Seizure disorder on medications
* HIV positive status
* Known major fetal anomalies
* Multifetal gestation

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 220 (Actual)
Dates: Start 2019-05-06 (Actual); Primary Completion 2023-04-10 (Actual); Study Completion 2023-04-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: farah Amro, MD, Principal Investigator — University of Texas Health Science Center of Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 162 mg/Day Aspirin | 81 mg/Day Aspirin
Started | 110 | 110
Completed | 107 | 102
Not Completed | 3 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 162 mg/Day Aspirin | 81 mg/Day Aspirin | Total
Number analyzed (Participants) | 110 | 110 | 220
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 30 [26 to 34] | 29 [25 to 33] | 29 [25 to 34]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 110 | 110 | 220
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African American | 52 | 59 | 111
  Hispanic/Latina | 34 | 25 | 59
  White | 8 | 7 | 15
  Unknown or not reported | 16 | 19 | 35
Region of Enrollment [Number; unit: participants]
  United States | 110 | 110 | 220
Insurance Type [Count of Participants; unit: Participants]
  Private | 10 | 11 | 21
  Government assisted (Medicaid, Medicare or other federal or state funded assistance program) | 99 | 99 | 198
  Self pay | 1 | 0 | 1
Gestational age at enrollment [Median (Inter-Quartile Range); unit: weeks] | 15.9 [13.6 to 17.6] | 15.6 [13.6 to 17.7] | 15.64 [13.57 to 17.71]
Body Mass Index [Median (Inter-Quartile Range); unit: kg/m^2] | 37 [33 to 43] | 38 [34 to 44] | 37.88 [33.60 to 43.73]
Number of Participants who are Nulliparous [Count of Participants; unit: Participants] | 19 | 27 | 46
Number of Participants with Systemic Lupus Erythematosus [Count of Participants; unit: Participants] | 2 | 1 | 3
Number of Participants who use tobacco during pregnancy [Count of Participants; unit: Participants] | 2 | 1 | 3
History of preeclampsia in prior pregnancy [Count of Participants; unit: Participants] | 37 | 30 | 67
Number of participants with Type 1 diabetes [Count of Participants; unit: Participants] | 3 | 5 | 8
Number of participants with type 2 diabetes [Count of Participants; unit: Participants] | 41 | 43 | 84
Number of participants diagnosed with gestational diabetes before 20 weeks [Count of Participants; unit: Participants] | 3 | 7 | 10
Number of participants enrolled prior to 16 weeks [Count of Participants; unit: Participants] | 55 | 58 | 113
Number of participants on aspirin prior to enrollment [Count of Participants; unit: Participants] | 23 | 21 | 44

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Preeclampsia Diagnosis With Severe Features Based on Clinician Diagnosis
Description: based on American College Obstetrics and Gynecology (ACOG) guidelines
Time Frame: 3-7 months
Measure: Count of Participants; unit: Participants
Arm/Group | 162 mg/Day Aspirin | 81 mg/Day Aspirin
Number analyzed (Participants) | 107 | 102
Participants | 37 | 41

2. Secondary Outcome: Maternal Outcomes- Number of Participants Who Delivered Due to Preeclampsia With Severe Features
Time Frame: less than 37 weeks gestational age (GA)
Measure: Count of Participants; unit: Participants
Arm/Group | 162 mg/Day Aspirin | 81 mg/Day Aspirin
Number analyzed (Participants) | 107 | 102
Participants | 22 | 21

3. Secondary Outcome: Maternal Outcomes-Number of Participants With Gestational Hypertension
Description: development of hypertension anytime during pregnancy based on ACOG guidelines
Time Frame: 3-7 months
Measure: Count of Participants; unit: Participants
Arm/Group | 162 mg/Day Aspirin | 81 mg/Day Aspirin
Number analyzed (Participants) | 107 | 102
Participants | 13 | 20

4. Secondary Outcome: Maternal Outcomes- Number of Participants With Placenta Abruption
Description: Placental abruption occurs when the placenta separates from the inner wall of the uterus before birth. As assessed by treating OBGYN
Time Frame: 1 day
Measure: Count of Participants; unit: Participants
Arm/Group | 162 mg/Day Aspirin | 81 mg/Day Aspirin
Number analyzed (Participants) | 107 | 102
Participants | 3 | 3

5. Secondary Outcome: Maternal Outcomes- Number of Participants With Eclampsia
Description: onset of seizures (convulsions) in a woman with pre-eclampsia per ACOG guidelines
Time Frame: 20 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | 162 mg/Day Aspirin | 81 mg/Day Aspirin
Number analyzed (Participants) | 107 | 102
Participants | 0 | 0

6. Secondary Outcome: Maternal Outcomes- Number of Participants With HELLP Syndrome
Description: group of symptoms that occur in pregnant women who have: hemolysis(H): (the breakdown of red blood cells)elevated liver enzymes (EL). low platelet (LP) count. Assessed by ACOG guidelines and measured in urine and blood samples
Time Frame: 4 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | 162 mg/Day Aspirin | 81 mg/Day Aspirin
Number analyzed (Participants) | 107 | 102
Participants | 0 | 0

7. Secondary Outcome: Maternal Outcomes- Number of Participants With Postpartum Hemorrhage
Description: excessive bleeding following the birth of a baby
Time Frame: 1-24 hrs post delivery
Measure: Count of Participants; unit: Participants
Arm/Group | 162 mg/Day Aspirin | 81 mg/Day Aspirin
Number analyzed (Participants) | 107 | 102
Participants | 11 | 9

8. Secondary Outcome: Maternal Outcomes- Number of Participants With Other Maternal Bleeding
Description: any other bleeding associated with birth not otherwise categorized
Time Frame: during labor to 24 hrs post delivery
Measure: Count of Participants; unit: Participants
Arm/Group | 162 mg/Day Aspirin | 81 mg/Day Aspirin
Number analyzed (Participants) | 107 | 102
Participants | 0 | 0

9. Secondary Outcome: Maternal Outcomes- Number of Participants That Required Blood Transfusion
Description: peripartum
Time Frame: during delivery
Measure: Count of Participants; unit: Participants
Arm/Group | 162 mg/Day Aspirin | 81 mg/Day Aspirin
Number analyzed (Participants) | 107 | 102
Participants | 8 | 6

10. Secondary Outcome: Neonatal Outcome- Gestational Age at Delivery
Time Frame: at delivery
Measure: Median (Inter-Quartile Range); unit: weeks
Arm/Group | 162 mg/Day Aspirin | 81 mg/Day Aspirin
Number analyzed (Participants) | 107 | 102
weeks | 36.30 [34.40 to 37.40] | 37.20 [35.10 to 38.20]

11. Secondary Outcome: Neonatal Outcomes-Delivery at < 37 Weeks
Time Frame: at delivery
Measure: Count of Participants; unit: Participants
Arm/Group | 162 mg/Day Aspirin | 81 mg/Day Aspirin
Number analyzed (Participants) | 107 | 102
Participants | 58 | 45

12. Secondary Outcome: Neonatal Outcomes-Apgar Score < 5 at 5 Minutes
Description: The Apgar score is determined by evaluating the newborn baby on each of five criteria (appearance, pulse, grimace, activity, respiration) on a scale from zero to two, then summing the five values obtained. The total score ranges from zero to 10. A higher score indicates a better outcome.
Time Frame: 5 minutes post delivery
Measure: Count of Participants; unit: Participants
Arm/Group | 162 mg/Day Aspirin | 81 mg/Day Aspirin
Number analyzed (Participants) | 107 | 102
Participants | 4 | 3

13. Secondary Outcome: Neonatal Outcome-Small for Gestational Age
Description: Small for gestational age (SGA) means that a fetus or an infant is smaller or less developed than normal for the baby's sex and gestational age. Small for gestational age (SGA) is defined as a birth weight that is below the 10th percentile.
Time Frame: at delivery
Measure: Count of Participants; unit: Participants
Arm/Group | 162 mg/Day Aspirin | 81 mg/Day Aspirin
Number analyzed (Participants) | 107 | 102
Participants | 7 | 3

14. Secondary Outcome: Neonatal Outcome-Neonatal Intensive Care Unit (NICU) Length of Stay
Time Frame: from birth until discharge from NICU (about 1 to 4 weeks)
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | 162 mg/Day Aspirin | 81 mg/Day Aspirin
Number analyzed (Participants) | 107 | 102
days | 10 [4 to 17] | 10.5 [3.75 to 21.5]

15. Secondary Outcome: Neonatal Outcome- Number of Participants With Intraventricular Hemorrhage Grade III-IV
Description: bleeding inside or around the ventricles in the brain.
Time Frame: from birth until discharge from NICU (about 1 to 4 weeks)
Measure: Count of Participants; unit: Participants
Arm/Group | 162 mg/Day Aspirin | 81 mg/Day Aspirin
Number analyzed (Participants) | 107 | 102
Participants | 0 | 0

16. Secondary Outcome: Neonatal Outcome-Number of Participants With Bronchopulmonary Dysplasia
Description: chronic lung disease that affects newborns (mostly premature) and infants.
Time Frame: from birth until discharge from NICU (about 1 to 4 weeks)
Measure: Count of Participants; unit: Participants
Arm/Group | 162 mg/Day Aspirin | 81 mg/Day Aspirin
Number analyzed (Participants) | 107 | 102
Participants | 0 | 0

17. Secondary Outcome: Neonatal Outcome-Number of Participants With Necrotizing Enterocolitis
Description: medical condition where a portion of the bowel dies
Time Frame: from birth until discharge from NICU (about 1 to 4 weeks)
Measure: Count of Participants; unit: Participants
Arm/Group | 162 mg/Day Aspirin | 81 mg/Day Aspirin
Number analyzed (Participants) | 107 | 102
Participants | 1 | 0

ADVERSE EVENTS:
Time Frame: From enrollment (12 to 20.6 weeks gestational age) to 6 weeks post-partum
Arm/Group | 162 mg/Day Aspirin | 81 mg/Day Aspirin
All-Cause Mortality (participants affected / at risk) | 0/110 | 0/110
Serious Adverse Events (participants affected / at risk) | 24/110 | 19/110
Other Adverse Events (participants affected / at risk) | 51/110 | 61/110
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 162 mg/Day Aspirin (N=110) | 81 mg/Day Aspirin (N=110)
Placenta Abruption (Pregnancy, puerperium and perinatal conditions) | 3 | 3
Postpartum hemorrhage (Pregnancy, puerperium and perinatal conditions) | 11 | 9
Maternal blood transfusion (Pregnancy, puerperium and perinatal conditions) | 8 | 6
Fetal Heart Defect (Congenital, familial and genetic disorders) | 2 | 0
Kidney Malformation (Congenital, familial and genetic disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 162 mg/Day Aspirin (N=110) | 81 mg/Day Aspirin (N=110)
Preeclampsia (Pregnancy, puerperium and perinatal conditions) | 37 | 41
Gestational hypertension (Pregnancy, puerperium and perinatal conditions) | 13 | 20
Necrotizing Enterocolitis (Gastrointestinal disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-03-08): https://cdn.clinicaltrials.gov/large-docs/60/NCT03961360/Prot_SAP_000.pdf